CLINICAL TRIAL: NCT01981161
Title: Essai de Phase IV, Multicentrique, Ouvert, Visant à Tester la différence d'efficacité du Natalizumab, Versus le Fingolimod, 2 médicaments Ayant Une AMM Pour le Traitement de la sclérose en Plaques
Brief Title: Difference in Efficacy of Natalizumab Versus Fingolimod for the Treatment of Multiple Sclerosis
Acronym: BEST-MS
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: 1235207
Record Dates: First submitted 2013-11-04; First posted 2013-11-11 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Multiple Sclerosis
Keywords: progressive multifocal leucoencephalopathy; JC virus; Zoster infection
MeSH Terms: conditions — Multiple Sclerosis; Leukoencephalopathy, Progressive Multifocal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine and blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Fingolimod: patients treated by Fingolimod will have biological samples and clinical data
  Interventions: Procedure: biological samples and clinical data
- Natalizumab: patients treated by Natalizumab will have biological samples and clinical data
  Interventions: Procedure: biological samples and clinical data

INTERVENTIONS:
Procedure: biological samples and clinical data

SUMMARY:
Under the escalation treatment strategy when a patient displays breakthrough disease parameters under first line therapy, MS physicians are allowed by the EMEA to switch for Natalizumab (NTZ) or fingolimod (FGL). NTZ and FGL efficacy have been demonstrated by randomized therapeutic trial. As both treatments have been tested versus placebo a common way to compare them is to look at their respective annualized relapse risk ratio decrease. Roughly NTZ decrease by 70% and FGL by 50%. Nevertheless it is a terrible comparison since the placebo group had different behaviour in the 2 trials and the patients demographic features at baseline are also different. Therefore, it is right now totally impossible to compare these 2 drugs with a decent methodology. Only a head-to-head comparison could do it. Unfortunately this head-to-head comparison is not available and will not probably be done under the drug companies initiative. During the time of this study, we will perform a phase IV, observational, prospective head-to-head comparison of NTZ versus FGL efficacy in 600 patients. Our primary end point will be disease free patients after 1 year of treatment. Further, this trial will allow us to collect new biological samples, useful for a validation our project main aim. Further these new samples will be obtained from 3 European countries, which is a must if we want to generalize our conclusion obtained from a French cohort. Cooperation at the European level is thus essential for the implementation of this project .

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of relapsing-remitting MS in line with McDonald criteria;
* patient needing to be treated with FGL or NTZ, either:

  * Patients who have not responded to complete and well-conducted treatment with beta interferon. The patients should have presented at least one relapse during the course of the previous year while they were receiving treatment, and should present at least 9 hyper-intense lesions within T2 on a cerebral MRI, or at least 1 enhancing lesion following injection of Gadolinium; or
  * Patients presenting severe and rapidly developing relapsing-remitting multiple sclerosis, defined by 2 debilitating relapses or more during the course of one year, combined with 1 or more high-intensity lesion(s) following injection of Gadolinium on a cerebral MRI, or a significant increase in lesion load within T2 compared to a recent prior MRI.
* EDSS score between 0 and 6, not inclusive;
* patient who give informed consent, and signed the consent form;
* patient available for 12-month follow-up.

Exclusion Criteria:

* General exclusion criteria: The patient is subject to judicial protection, supervision or guardianship, the patient is pregnant, is about to give birth, or is breast-feeding, or there is an existing medical or major psychiatric condition that, in the investigator's opinion, could represent a risk for the subject or could compromise compliance with the study protocol.
* Contraindication to the use of NTZ and FGL in line with the marketing authorisation: for NTZ, the risk of tuberculosis assessed by means of intracutaneous reaction or quantiferon dosage, for FGL, positive VZV serology and an absence of risk factors for bradycardia and heart rate problems, and for both molecules, an absence of biological signs suggesting immunodepression (negative HIV serology, normal CD3, CD4, CD8 and CD19 levels, weight-adjusted dosage of immunoglobulin normal).
* prior treatment with FGL or NTZ;
* prior treatment with Mitoxantrone or Cyclophosphamide type immunosuppressants during the 5 years before inclusion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2013-11-19 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Disease free patients | 1 year

SECONDARY OUTCOMES:
comparing the efficacy of Natalizumab with that of Fingolimod with regard to the annual incidence rate (comparison against the annual incidence rate criterion after 1 year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David Brassat, MD,PHD, Principal Investigator — U H Toulouse
Locations (12):
- France (10):
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHU Caen, Caen
  - Chu Lille, Lille
  - Chu La Timone, Marseille
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - CHU Nîmes, Nîmes
  - CHRU Strasbourg, Strasbourg
- Université de Muenter, Münster, Germany
- Hôpital Vall D'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided